CLINICAL TRIAL: NCT06034639
Title: AI Based Multi-modal Parameter of Peripheral Blood Cells (MMPBC) Predicts Survival Risk in Critically Ill Children: a Multicenter, Retrospective Cohort Study
Brief Title: AI Based Multi-modal Parameter of Peripheral Blood Cells (MMPBC) Predicts Survival Risk in Critically Ill Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Hongwei Zhou, high professional title, Zhujiang Hospital
Other Study IDs: GPCRCLM0001
Record Dates: First submitted 2023-08-11; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Children
Keywords: artificial Intelligence; critically ill children; survival Risk

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: No Intervention

SUMMARY:
This study aims to investigate whether an AI prediction model based on blood cell multi-modal data can achieve early warning of survival risk in critically ill children through a large-scale multi-center cohort of critically ill children.

DETAILED DESCRIPTION:
According to the definition of the United Nations Children's Fund (UNICEF), children are individuals between the ages of 0 and 18. Critically ill children are those who are admitted to the PICU or NICU and suffer from severe illnesses that require special treatment. These illnesses may endanger the child's life. Studies have reported that the international PICU mortality rate in developed countries is 2% to 3%; in recent years, the in-hospital mortality rate of PICU in China is 4.7% to 6.8%. The assessment of the survival risk of critically ill children has always been a focus of attention. Traditional assessment methods include physiological indicators, scoring tools, severity of illness, and diagnosis time, which can help doctors make decisions to a certain extent, but their predictive ability is limited and difficult to comprehensively reflect the child's physiological status and disease progression.

With the development of technology and social progress, blood cell analysis is evolving towards a highly integrated platform of multiple cell analysis technologies that provide more accurate results, more comprehensive parameters, and faster detection. Cell analysis applications are increasingly focused on the identification and alarm capabilities of abnormal samples, including reticulocytes, nucleated red blood cells, and immature granulocytes. In 2009, Mindray Group, in collaboration with the National Key Laboratory of Fine Chemicals, developed a new nucleic acid-targeted fluorescent dye that meets the requirements of blood cell analysis (the patented fluorescent dye won the National Science and Technology Progress Second Prize). This breakthrough technology overcame international intellectual property barriers and developed the first high-end blood cell analyzer, the BC-6800, with functions to detect nucleated red blood cells and reticulocytes. The device has been successfully promoted to over 90% of tertiary hospitals in China. While detecting routine blood cell ratios, this blood cell analyzer actually generates a large amount of multi-modal data on cell distribution characteristics, including cell distribution width and abnormal cell ratios. However, so far, these multi-modal data have not been fully utilized in clinical practice.

Preliminary exploration of multi-modal cell data has demonstrated its enormous value in predicting, diagnosing, and prognosing infectious diseases in small populations. This study aims to retrospectively collect clinical data and blood cell multi-modal data from NICU and PICU hospitalized children in multiple centers across China, to establish a national multi-center blood cell multi-modal database with no less than 100,000 people, and to use artificial intelligence technology to achieve accurate, repeatable, and unbiased identification and classification based on differences in cell morphology and structural distribution. A high-performance prediction model will be constructed in the discovery cohort to predict the survival risk of critically ill children; the performance of the model will be validated in the validation cohort to evaluate its applicability in the Chinese population of critically ill children. This study will provide solid evidence for evidence-based medicine based on multi-center cohort studies and offer potential new inspection technologies for predicting the survival risk of critically ill children, providing auxiliary decision support for clinicians, improving the survival rate of critically ill children, and promoting the development of precision medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Children who were admitted to NICU and PICU from January 1, 2018, to March 31, 2023.
2. Age <18 years, gender not limited.
3. Blood routine tests were performed using Mindray Medical's five-category blood cell analyzer (including BC6000, BC6000PLUS, BC6800PLUS, and BC7500 series), and the instrument or computer system retained relatively complete blood cell multi-modal data.
4. Detailed clinical medical records related to this study can be obtained.
5. Patients who were repeatedly admitted to NICU or PICU and had different conditions, causes, and outcomes each time were counted as new cases.

Exclusion Criteria:

1. Children with congenital immunodeficiency.
2. Children with blood diseases, including iron-deficiency anemia, macrocytic anemia, hereditary spherocytosis, glucose-6-phosphate dehydrogenase deficiency, thalassemia, autoimmune hemolytic anemia, aplastic anemia, immune thrombocytopenia, acute lymphoblastic leukemia, acute non-lymphoblastic leukemia, multiple myeloma, allergic purpura, myelodysplastic syndrome, etc.
3. Children with genetic metabolic diseases, including galactosemia, mucopolysaccharidosis, glycogen storage disease, phenylketonuria, albinism, alkaptonuria, hypoxanthine-guanine phosphoribosyltransferase deficiency, chromhidrosis, Goucher disease, Tay-Sachs disease, etc.
4. Children with chromosomal diseases, including Down syndrome, trisomy 18, etc.
5. Children who received blood products within six months, including transfused blood components, human immunoglobulin, etc.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The included population in this study consists of children who meet the following criteria: they were admitted to NICU and PICU between January 1, 2018, and March 31, 2023, and are under the age of 18 with no gender limitation. These children underwent blood routine tests using Mindray Medical's five-category blood cell analyzer, and the instrument or computer system retained relatively complete blood cell multi-modal data. Additionally, they have detailed clinical medical records related to this study. Excluded from the study are children with underlying blood, genetic, or chromosomal diseases, those who have received blood products in the past six months, and non-critically ill children who temporarily stayed in NICU or PICU due to bed availability issues in other wards.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
death | through study completion, an average of 1 month
  diagnosis time based on medical records
multiple organ dysfunction syndrome(MODS) | through study completion, an average of 1 month
  diagnosis time based on medical records
sepsis | through study completion, an average of 1 month
  diagnosis time based on medical records

SECONDARY OUTCOMES:
disseminated intravascular coagulation(DIC) | through study completion, an average of 1 month
  diagnosis time based on medical records
chronic lung disease or acute respiratory distress syndrome | through study completion, an average of 1 month
  diagnosis time based on medical records
shock | through study completion, an average of 1 month
  diagnosis time based on medical records
Length of stay in the pediatric intensive care unit(PICU) or neonatal intensive care unit(NICU) hospitalization duration | through study completion, an average of 1 month
  diagnosis time based on medical records
brain injury or neurological complications | through study completion, an average of 1 month
  diagnosis time based on medical records

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China